CLINICAL TRIAL: NCT02878005
Title: A Prospective and Randomized Study Comparing the New Intubating Laryngeal Tube Suction and the Ambu AuraGain in Adult Patients
Brief Title: A Comparison Between the Intubating Laryngeal Tube Suction and the Ambu AuraGain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS.GAITINI, M.D., Bnai Zion Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-LG-005
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Intubation; Difficult
Keywords: Intubating Laryngeal Tube; blind intubation; fiberoptic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubating laryngeal Tube Suction (Active Comparator): Intubating laryngeal Tube Suction
  Interventions: Device: Intubating Laryngeal Tube Suction; Device: Ambu AuraGain Laryngeal Mask
- Ambu AuraGain Laryngeal Mask (Active Comparator): Ambu AuraGain Laryngeal Mask
  Interventions: Device: Intubating Laryngeal Tube Suction; Device: Ambu AuraGain Laryngeal Mask

INTERVENTIONS:
Device: Intubating Laryngeal Tube Suction — Intubating Laryngeal Tube Suction
Device: Ambu AuraGain Laryngeal Mask — Ambu AuraGain Laryngeal Mask

SUMMARY:
The intubating Laryngeal Tube Suction-Disposable is a new version of the Laryngeal Tube-Suction. It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube either blindly or with fiberoptic guidance.This study was designed to assess the success rate of blind and fiberoptic endotracheal intubation using iLTS-D, in comparison with the and Ambu® AuraGain™ in adult patients.

DETAILED DESCRIPTION:
The intubating Laryngeal Tube Suction-Disposable (iLTS-D) (VBM Medizintechnik GmbH, Sulz, Germany) is a new updated version of the Laryngeal Tube-Suction Disposable (LTS-D) It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube (ETT) either blindly or with fiberoptic guidance. Similarly As in to the LTS-D, the iLTS-D also has a separate channel for the purpose of placement of gastric tubes placement up to a size of 18 Fr.

The iLTS-D comes in one size. According to the depth of insertion, this device is equivalent to size 4 for patients 175patients 175 to 190 cm tall, or size 5 for patients taller than 190 cm. The iLTS-D is provided by the manufacturer with a compatible 7.5mm ETT and with a plastic stabilizer for removal of the device.

The current randomized study was designed to assess the success rate of blind and fiberoptic endotracheal intubation using iLTS-D, in comparison with the and Ambu® AuraGain™ in adult patients under general anesthesia

ELIGIBILITY:
Inclusion Criteria:

American Society Anesthesiology I and II

Exclusion Criteria:

Difficult intubation, Cervical pathology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time to performe blind intubation measure in second | 30 seconds

SECONDARY OUTCOMES:
Time to performe fiberoptic intubation in second | 60 seconds

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Somri M, Hochman O, Gaitini L, Hossein J, Gomez-Rios MA. The intubating laryngeal tube (iLTS-D) versus Ambu(R) Auragain as a conduit facilitating fiberoptic tracheal intubation in adult population: results from a prospective randomized controlled trial. Minerva Anestesiol. 2022 Dec;88(12):1074-1076. doi: 10.23736/S0375-9393.22.16731-3. No abstract available. PMID 36445250